CLINICAL TRIAL: NCT00603356
Title: A Phase 1 Dose Escalation Study of Daily Oral OSI-930 and Erlotinib (Tarceva) in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of OSI-930 and Erlotinib in Cancer Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-930-103
Record Dates: First submitted 2007-12-26; First posted 2008-01-29 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Solid Tumors
Keywords: GIST; Ovarian Cancer; Mesothelioma; Renal; Colorectal Cancer; Sarcoma; NSCLC; Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Mesothelioma; Colorectal Neoplasms; Sarcoma; Neoplasms | interventions — OSI 930; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Dose Escalation
  Interventions: Drug: OSI-930 and erlotinib

INTERVENTIONS:
Drug: OSI-930 and erlotinib — OSI-930 administered daily in combination with Erlotinib at increasing doses until disease progression or unacceptable toxicity

SUMMARY:
This is a Phase I, dose escalation, safety study of OSI-930 and Erlotinib in cancer tumors.

DETAILED DESCRIPTION:
Multicenter, open-label, phase 1, dose escalation study to determine the maximum tolerated dose of OSI-930 and Erlotinib.

Patients may continue to receive OSI-930 and Erlotinib until one of the following occurs: disease progression, adverse event requiring withdrawal, failure to recover from toxicity despite a 14-day dosing interruption, medical or ethical reasons, patient request, or patient death.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytologically documented malignancy that is now advanced and/or metastatic and refractory to established forms of therapy or for which no effective therapy exists
* Age greater than or equal to 18 years
* ECOG PS 0-2
* ANC greater than or equal to 1.5 x 10^9/L
* Bilirubin less than or equal to 1.5 x upper limit of normal (ULN), AST and ALT less than or equal to 2.5 x ULN
* Creatinine less than or equal to 1.5 ULN
* Predicted life expectancy greater than or equal to 12 weeks
* Prior chemotherapy is permitted provided that a minimum of 3 weeks has elapsed
* Prior tyrosine kinase inhibitor therapy is permitted
* Patients must have recovered from any treatment-related toxicities (with some exceptions) prior to registration
* Prior hormonal therapy is permitted provided it is discontinued prior to registration (with the exception of prostate cancer patients who have been on hormone therapy for at least 3 months)
* Prior radiation therapy is permitted provided that it did not exceed 25% of bone marrow reserve and patients have recovered from the toxic effects (a minimum of 21 days must have elapsed unless the radiotherapy was palliative and nonmyelosuppressive)
* Prior surgery is permitted, provided that wound healing has occurred prior to registration
* Patients must use proactive effective contraceptive measures throughout the study
* Provide written informed consent
* Accessible for repeat dosing and follow-up
* Adequate hematopoietic, hepatic, and renal function

Exclusion Criteria:

* Significant cardiac disease unless well controlled
* Current or former smokers, unless patients stopped smoking greater than 3 months prior to registration
* Active or uncontrolled infections of serious illnesses or medical conditions that could interfere with participation
* History of unacceptable toxicity with previous EGFR inhibitor therapy
* History of any psychiatric condition that might impair the patient's ability to provide informed consent or participate
* Use of CYP3A4 inducers/inhibitors during the 14 days prior to first dose
* Pregnant or breast-feeding females
* Symptomatic brain metastases which are not stable, require steroids, are potentially life-threatening or that have required radiation within the last 28 days
* History of allergic reaction attributed to a similar compound as study drug
* GI abnormalities including inability to take oral medications, required for IV alimentation
* Clinically significant ophthalmologic abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD), evaluate the pharmacokinetic profiles | 18 months

SECONDARY OUTCOMES:
Safety, evaluate pharmacodynamic relationships | 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States
- The Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom